CLINICAL TRIAL: NCT01763268
Title: Immunogenicity and Reactogenicity of a Trivalent MMR (Trivivac) in Healthy Infants
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Sirikit National Institute of Child Health (Other Government)
Responsible Party: Principal Investigator, Warunee Punpanich Vandepitte, Assistant Professor, Dr., Queen Sirikit National Institute of Child Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Trivivac2012
Record Dates: First submitted 2013-01-03; First posted 2013-01-08 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Immunogenicity; Reactogenicity
Keywords: Immunogenicity; Reactogenicity; Trivivac; Measles; Mump; Rubella
MeSH Terms: conditions — Measles; Rubella

ARMS (1):
- Trivivac (Experimental): Children who receive Trivivac vaccine
  Interventions: Biological: Trivivac vaccine

INTERVENTIONS:
Biological: Trivivac vaccine — Trivalent MMR vaccine

SUMMARY:
Open-label, single-arm trial, Primary Objectives included:

1. To assess the immunogenicity of TrivivacTM administered in healthy infants aged between 9-14 months.
2. To assess the safety (reactogenicity) of TrivivacTM administered in healthy infants aged between 9-14 months.

The study will be done on healthy infants, 9-14 months of age. After enrolment, the infants will be given one dose of primary vaccination MMR (TrivivacTM),SEVAPHARMA BiogenetechLtd. study vaccines will be administered subcutaneously into the anterolateral aspect of right thigh.outer aspect of the upper arm. Subjects will be followed at approximately 6 weeks after primary vaccination to evaluate response to primary immunization of this vaccine. Blood sample will be collected from subjects at visit 1 (prior to immunization) and visit 2 (6 weeksone month after completion of this first dose of immunization). The serum samples will be analysed for Anti-measles, Anti-mumps and Anti-rubella antibodies. Proportion of subjects achieving seroprotection and geometric mean titers of antibody against measles, mumps, rubella at 6 weeks after one dose vaccination of MMR vaccine at aged 9-14 months will be evaluated. Adverse reactions will be observed on each vaccination day (up to 30 minutes) and for 4 days (Day 0-3) after each dose. Adverse reactions will also be monitored for 30 days following each vaccination. Serious adverse events will be monitored for the entire study duration.

ELIGIBILITY:
Inclusion Criteria:

1. Infants aged 9-14 months whose parents/LAR give written informed consent prior to the study entry.
2. Infants with good health as determined by: Medical history, Physical examination, Clinical judgment of the investigator
3. Infants who are not seroprotected against MMR virus by virtue of previous immunization and/or proven prior infection.

Exclusion Criteria:

1. Children whom parents or LAR are unwilling or unable to give written informed consent to participate in the study.
2. Any evidence of acute illness or infection within past 14 days.
3. Planned or elective surgery during the course of the study.
4. Infants born before the 37th week of gestation.
5. Birth weight less than 2.5 kg.
6. Infants with a known or suspected impairment of the immune function, or those receiving immunosuppressive therapy, or having received immunosuppressive therapy within 1 month prior to study entry (including systemic corticosteroids) or those who have received a parenteral immunoglobulin preparation.
7. Any history suggestive of thrombocytopenia or a bleeding disorder.
8. Infants who have received any blood products (within 3 months prior to study entry), cytotoxic agents or radiotherapy.
9. Infants with history of anaphylaxis, or any serious vaccine reaction, or allergy to any vaccine component (e.g. neomycin, gelatine, canine proteins).
10. Infants with any serious chronic disease such as cardiac, autoimmune disease or insulin dependent diabetes or with any condition that in the opinion of the investigator might interfere with the evaluation of the study objectives.
11. Infants whose families are planning to leave the area of the study site before the end of the study period.

Ages: 9 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-01 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity as measured by the proportion of subjects achieving seroprotection against measles, mumps and rubella | 6 weeks after vaccination
  Immunogenicity of Trivivac vaccine is determined by proportion of subjects achieving seroprotection against measles, mumps and rubella at 6 weeks (42 days) after application of first dose of vaccine MMR. The amount of specific antibodies against measles, mumps and rubella will be evaluated in sera collected approximately 42+ 7 days following primary vaccination with the Trivivac vaccine.
  Seroconversion and GMT against measles, mumps, and rubella will be defined by Enzyme immunoassay for the qualitative detection and quantitative determination of specific IgG antibodies against measles, mumps and rubella virus in human serum (Enzygnost® Anti-Measles Virus/IgG, Anti-Mumps Virus/IgG and Anti-Rubella Virus/IgG; SIEMENS).

SECONDARY OUTCOMES:
Reactogenicity as measured by the prevalence of local and systemic adverese reaction | Day0 to day3 after vaccination
  Occurrence, intensity and relationship to vaccination of early expected and unexpected local and systemic adverse drug reactions reported during the 4-day (Day 0-3) follow-up period after vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Sirikit National Institute of Child Health, Bangkok, Bangkok, Thailand